CLINICAL TRIAL: NCT02675803
Title: A Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of VAY736 in Rheumatoid Arthritis Patients
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of VAY736 in Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVAY736X2101; 2010-020156-65
Record Dates: First submitted 2015-07-09; First posted 2016-02-05 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2019-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ianalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VAY736 (Experimental): VAY736 active
  Interventions: Biological: VAY736
- Placebo (Placebo Comparator): VAY736 placebo
  Interventions: Biological: VAY736 placebo

INTERVENTIONS:
Biological: VAY736 — VAY736 treatment
  Arms: VAY736
Biological: VAY736 placebo — VAY736 placebo
  Arms: Placebo

SUMMARY:
This study investigated the safety and tolerability of VAY736 administered as single ascending doses of intravenous infusion, subcutaneous injection and repeated subcutaneous injections in rheumatoid arthritis patients.

DETAILED DESCRIPTION:
This study had three sequential parts which investigated the safety and tolerability of VAY736 administered as single ascending doses of intravenous infusion (Part 1), single ascending doses of subcutaneous injection (Part 2), and repeated subcutaneous injections of fixed doses (Part 3), respectively, in rheumatoid arthritis patients. Part 1 was double blind, placebo controlled, with 11 cohorts. Part 2 was open-label study with 2 dosing cohorts. Part 3 was open-label study with 1 fixed-dose cohort.

ELIGIBILITY:
Inclusion Criteria:

* Active disease despite methotrexate treatment 5 to 20 mg/week for Parts 1 and 2; methotrexate treatment 5 to 20 mg/week for Part 3
* Fulfilled 2010 American College of Rheumatolody (ACR)/European League Against Rheumatism (EULAR) classification criteria for rheumatoid arthritis for Part 1 and Part 2. For Part 3, fulfilled 2010 American College of Rheumatolody (ACR)/)/European League Against Rheumatism (EULAR) classification criteria or/and 1987 American College of Rheumatolody (ACR) classification criteria for rheumatoid arthritis;
* Methotrexate ≥ 16 weeks, stable dose ≥ 8 weeks

Exclusion Criteria:

* Previous treatment with a B cell-depleting biologic agent.
* Autoimmune disease other than RA except concurrent Sjogren's syndrome
* Adult juvenile rheumatoid arthritis
* ARA functional class IV disease of ACR Revised Steinbrocker Classification

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-12-20 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by the number of patients wth adverse events | 27-188 weeks
  Part 1 The number of patients with adverse events after single intravenous (i.v.) dose of VAY736. Patients are assessed weekly up to 34 weeks post dose or until B cells reach the recovery criteria
  Part 2 The number of patients with adverse events after single subcutaneous (s.c.) dose of VAY736. Patients are assessed weekly, bi-weekly, then every 4, 8 and 12 weeks up to 188 weeks post dose or until B cells reach the recovery criteria.
  Part 3 The number of patients with adverse events after repeated subcutaneous (s.c) injections of a fixed dose of VAY736. Patients are assessed bi-weekly, then every 4 weeks and 8 weeks up to 27 weeks from the first dose.
Absolute bioavailability of VAY736: The ratio of area under curve (AUC) for s.c dose and for intravenous dose | 188 weeks
  Part 2 The ratio of area under curve (AUC) for single s.c dose and intravenous dose is determined
Plasma pharmacokinetics of VAY736: The area under the plasma concentration-time curve from time zero to the end of the dosing interval (AUCtau) | 27 weeks
  In Part 3:
  After the first and last s.c. doses, the area under the plasma concentration-time curve from time zero to the end of the dosing interval (AUCtau) will be determined
Plasma pharmacokinetics of VAY736: Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) | 27 weeks
  In Part 3:
  After the first and last s.c. doses, the Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) will be determined.
Plasma pharmacokinetics of VAY736: Observed maximum plasma concentration following drug administration (Cmax) | 27 weeks
  In Part 3:
  After the first and last s.c. doses, the Observed maximum plasma concentration following drug administration (Cmax) will be determined
Plasma pharmacokinetics of VAY736: Time to reach the maximum concentration after drug administration (Tmax) | 27 weeks
  In Part 3:
  After the first and last s.c. doses, the time to reach the maximum concentration after drug administration (Tmax) will be determined
Plasma pharmacokinetics of VAY736: The terminal elimination half-life (T1/2) | 27 weeks
  In Part 3:
  After the first and last s.c. doses, the terminal elimination half-life (T1/2) will be determined
Plasma pharmacokinetics of VAY736: Area under the plasma concentration-time curve from time zero to infinity (AUCinf) | 27 weeks
  In Part 3:
  After the first and last s.c. doses, Area under the plasma concentration-time curve from time zero to infinity (AUCinf) will be determined.
Plasma pharmacokinetics of VAY736: concentration of VAY736 during the treatment period, before each dose (Ctrough) | 27 weeks
  In Part 3:
  After the first and last s.c. doses, the concentration of VAY736 during the treatment period, before each dose (Ctrough) will be determined
Safety and tolerability as measured by the percentage of patients wth adverse events | 27-188 weeks
  Part 1 The percentage of patients with adverse events after single intravenous (i.v.) dose of VAY736. Patients are assessed weekly up to 34 weeks post dose or until B cells reach recovery criteria.
  Part 2 The percentage of patients with adverse events after single subcutaneous (s.c.) dose of VAY736. Patients are assessed weekly, bi-weekly, then every 4, 8 and 12 weeks up to 68 weeks post dose or until B cells reach recovery criteria..
  Part 3 The percentage of patients with adverse events after repeated subcutaneous (s.c) injections of a fixed dose of VAY736. Patients are assessed bi-weekly, then every 4 weeks and 8 weeks up to 27 weeks from the first dose.

SECONDARY OUTCOMES:
pharmacodynamics of VAY736 | 27-188 weeks
  B cell depletion/recovery after single i.v. dose of VAY736, single s.c. dose of VAY736 and multiple fixed s.c. doses of VAY736 administration in the 3 parts of the study
Immunogenicity of VAY736 | 27-188 weeks
  Immunogenicity after administration of single i.v. dose of VAY736, single s.c. dose of VAY736 and multiple fixed s.c. doses of VAY736 in 3 parts of the study.
Plasma bioavailability of VAY736: The ratio of area under curve (AUC) for repeated s.c doses and for intravenous dose | 27 weeks
  Part 3 The ratio of area under curve (AUC) for repeated s.c doses and for intravenous dose is determined
Plasma pharmacokinetics of VAY736: Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) | 34-188 weeks
  The area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) will be determined after single i.v. dose and s.c. dose of VAY736 in Part 1 and Part 2 respectively
Plasma pharmacokinetics of VAY736: Area under the plasma concentration-time curve from time zero to infinity (AUCinf) | 34-188 weeks
  The area under the plasma concentration-time curve from time zero to infinity (AUCinf) will be determined after single i.v. dose and s.c. dose of VAY736 in Part 1 and Part 2 respectively.
Plasma pharmacokinetics of VAY736: Observed maximum plasma concentration following drug Administration (Cmax) | 34-188 weeks
  The Observed maximum plasma concentration following drug administration (Cmax) will be determined after single i.v. dose and s.c. dose of VAY736 in Part 1 and Part 2 respectively
Plasma pharmacokinetics of VAY736: Time to reach the maximum concentration after drug administration (Tmax) | 34-188 weeks
  The time to reach the maximum concentration after drug administration (Tmax) will be determined after single i.v. dose and s.c. dose of VAY736 in Part 1 and Part 2 respectively

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CVAY736X2101 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17297
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=422